CLINICAL TRIAL: NCT06319001
Title: Cardiovascular Reactivity to Physical Stress: Strategies and Mechanisms
Brief Title: Cardiovascular Reactivity to Physical Stress
Acronym: REACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Ann-Katrin Grotle, Associate professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2688791
Record Dates: First submitted 2024-02-11; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Blood Pressure; Stress, Physiological
Keywords: Cardiovascular reactivity; Neural control of blood pressure; Metaboreflex; Cold pressor response

STUDY DESIGN:
Intervention Model Description: Combined randomized controlled trial with two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive stress education (PSE) (Experimental): This intervention will consist of standardized information about the relationships between expectations and the stress response. Using the CATS as a theoretical framework, the participants will be explained that when people face stressors, i.e., pain, heat, and cold water, the expectations about handling the situation will influence both the experience (e.g., pain) and the physiological stress response.
  Interventions: Other: Low-volume high intensity exercise; Other: Combined intermittent sauna and cold water bath (sauna+cold bath).
- Neutral control (Sham Comparator): To control for the PSE intervention, the participants will receive 15 min of neutral information about the effects of physical exercise on cardiovascular fitness.
  Interventions: Other: Low-volume high intensity exercise; Other: Combined intermittent sauna and cold water bath (sauna+cold bath).

INTERVENTIONS:
Other: Low-volume high intensity exercise — This intervention will consist of 10 x 10-second interval sprints on a stationary bicycle interspersed with 50-second breaks between repetitions. The cycle resistance will be adjusted to the level equaling the highest power output, which will be determined during warm-up sprints.
Other: Combined intermittent sauna and cold water bath (sauna+cold bath). — This intervention will consist of 3x10 min bouts in the dry sauna interspersed with 2x 60 seconds of cold water immersion up to the neck.

SUMMARY:
It is well-accepted that an exaggerated blood pressure (BP) response to physical stress has a prognostic value, indicating a higher cardiovascular risk (e.g., sudden cardiac death, myocardial infarction, future hypertension, and left ventricular hypertrophy). However, there is a limited understanding of the underlying mechanisms and therapuetic strategies modulating this response. Therefore, this pilot project aims to explore whether one session of low-volume high-intensity interval training (low-volume HIIT) or combined intermittent heat and cold bath (sauna+cold bath) can decrease BP responses to physical stress. Furthermore, the secondary goal is to investigate whether one brief session learning about positive stress expectations magnifies the decrease in BP following low-volume HIIT and sauna+ cold bath.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 to 50 years
* Non-smoker.
* Non-obese (<30 kg/m2).
* Able to walk on a treadmill and cycle on a stationary bike without problems.
* No or little (frequency < 2 times per month) experience swimming with sauna and cold water.
* Proficient in Norwegian and able to provide informed consent.

Exclusion Criteria:

* Current or previous regular smoker
* Addictions to alcohol or illegal drugs
* Diagnosed with cardiovascular, respiratory, metabolic, or autoimmune diseases
* Taking prescription medication with known cardiovascular effects
* Judgment by a medical provider that exercise, heat therapy, or hydrotherapy poses an undue burden or risk.
* Cognitive or psychiatric impairment
* Lack of proficiency in Norwegian language oral or writing skills that will hamper the ability to participate in the interventions and fill out questionnaires.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (unit: mmHg) response to laboratory stressors | Assessment will be completed before intervention and approximately 30 minutes after intervention
  Response will be calculated as the change from baseline to peak. Stressors employed include handgrip exercise, post-exercise ischemia, and cold pressor test.

SECONDARY OUTCOMES:
Resting blood pressure (mmHg). | Assessment will be completed before intervention and approximately 30 minutes after intervention
Endothelial function (% dilation) | Assessment will be completed before intervention and approximately 30 minutes after intervention.
  Endothelial function will be assessed using the flow-mediated dilation technique following current guidelines.
Subjective ratings of expectancies (point score). | Assessment will be completed before intervention and approximately 30 minutes after intervention.
  Stress, pain, heat, and cold response expectancies will be assessed with single questions specifically targeted to the interventions and experimental tests using a Numeric Rating Scale (NRS) ranging from 0 = no stress, no pain, no discomfort (heat, cold) at all to 10 = worst possible pain, stress, heat/cold discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Vestland, Norway